CLINICAL TRIAL: NCT03578796
Title: Cognitive Impairment in ALS: Screening Tools, Experiences and Prognosis
Brief Title: Edinburgh Cognitive and Behavioural Amyotrophic Lateral Sclerosis Screen in Norway: A Prospective Cohort Study
Status: Active, not recruiting | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Collaborators: Western Norway University of Applied Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/2187-1
Record Dates: First submitted 2018-06-01; First posted 2018-07-06 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Amyotrophic Lateral Sclerosis; Cognitive Impairment
Keywords: Amyotrophic Lateral Sclerosis; Cognitive; Predictor
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Cognitive Dysfunction | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Persons with ALS: Persons With possible ALS-specific cognitive impairment will be tested With ECAS-N, MoCA, CDR and a questionnaire at 4 months (baseline) and 8 months (1. follow-up). Further evaluation will be with the questionnaire and CDR at each follow-up until 3 years or use of permanent ventilation support or Death. Information about use of advanced life-prolonging therapy will be collected from patient journal.
  Interventions: Diagnostic Test: ECAS-N; Diagnostic Test: MoCA; Diagnostic Test: CDR; Other: Questionnaire

INTERVENTIONS:
Diagnostic Test: ECAS-N — assessing ALS-specific cognitive impairment
  Other Names: Edinburgh cognitive and behavioural ALS screen
Diagnostic Test: MoCA — assessing cognitive impairment
  Other Names: Montreal cognitive assessment
Diagnostic Test: CDR — assessing global cognitive impairment, as well as possible diagnosis- and Level of dementia
  Other Names: Clinical dementia rating
Other: Questionnaire — Questions related to work situation and car driving

SUMMARY:
This study evaluate use of a translated Norwegian version of the Edinburgh cognitive and behavioral amyotrophic lateral sclerosis screen (ECAS-N) as an early predictor in car-driving, working and use of advanced life-prolonging therapy.

DETAILED DESCRIPTION:
Cognitive impairment is present in about 30-50% of the patients with amyotrophic lateral sclerosis (ALS). Screening of cognitive and behavioral impairment is a distinct recommendation in ALS-specific health care. However, knowledge in how cognitive impairment shall influence health-care professionals' information given to patients and in decision making is lacking.

One of the major challenges in ALS management is the decision-making on advanced therapy. There is a lack of knowledge in how cognitive impairment in ALS shall be interfere on complex medical treatment that will affect quality of life or life itself. This means significant implications not only to the ALS patient and the community, but also the family and especially the spouse. Thus, further investigation of the ECAS-N and its potential in clinical use is needed. The scale may contribute a more proactive treatment better tailored to individual needs. The objective is to evaluate if the ECAS-N can be applied as an early predictor in car-driving, working and use of advanced life-prolonging therapy

ELIGIBILITY:
Inclusion Criteria:

* Voluntary informed consent
* Native Norwegian speaker

Exclusion Criteria:

* Great difficulties in writing or reading
* Comorbid medical history
* Neurological disorders others than ALS
* Psychiatric history of importance to cognitive function

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who fullfill the inclusion criteria and attending to the ALS-clinic at HUH within 4 months after being diagnosed with ALS.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Dementia Rating (CDR) | 8 months
  We will use the total CDR score (minimum score = 0, maximum score = 18). Low scores indicate less problems than high scores.

SECONDARY OUTCOMES:
Clinical Dementia Rating (CDR) | 4 months
  We will use the total CDR score (minimum score = 0, maximum score = 18). Low scores indicate less problems than high scores.
Clinical Dementia Rating (CDR) | 3 years or until death
  We will use the total CDR score (minimum score = 0, maximum score = 18). Low scores indicate less problems than high scores.
Ability in car-driving | 8 months
  We will use a categorical variable (yes or no) and time of change to reduced function.
Ability in car-driving | 4 months
  We will use a categorical variable (yes or no) and time of change to reduced function.
Ability in car-driving | 3 years or until death
  We will use a categorical variable (yes or no) and time of change to reduced function.
Working ability | 8 months
  We will use a categorical variable (yes or no) and time of change to reduced function.
Working ability | 4 months
  We will use a categorical variable (yes or no) and time of change to reduced function.
Working ability | 3 years or until death
  We will use a categorical variable (yes or no) and time of change to reduced function.
Use of Advanced life-prolonging therapy | 8 months
  We will use a categorical variable (yes or no) and time of change to reduced function.
Use of Advanced life-prolonging therapy | 4 months
  We will use a categorical variable (yes or no) and time of change to reduced function.
Use of Advanced life-prolonging therapy | 3 years or until death
  We will use a categorical variable (yes or no) and time of change to reduced function.

OTHER OUTCOMES:
Edinburgh cognitive and behavioral amyotrophic lateral sclerosis screen-Norwegian Version (ECAS-N) | 4 months
  We will use the ALS-specific sub-score (minimum score = 0, maximum score = 100), the ALS non-specific sub-score (minimum score = 0, maximum score = 36), a summed total ECAS-N score (minimum score =0, maximum score =136), the sub score of behavioural changes (minimum score = 0, maximum score = 10) and the sub score of psychotic change (minimum score = 0, maximum score = 3). A dichotomized cut-off scores for normality will also be used for the ALS-specific cut-off score of 65 or over, the non ALS-specific cut-off score of 24 or over and the total ECAS-N cut-off score of 92 or over. For the ALS-specific scores, non ALS-specific scores and total ECAS-N scores, high scores indicate less problems than low scores. For the sub score of behavioural change and the sub score of psychotic change, high scores indicate more problems than low scores.
Change from 4 months Edinburgh cognitive and behavioral amyotrophic lateral sclerosis screen-Norwegian Version (ECAS-N) at 8 months | 8 months
  We will use the changed ALS-specific sub-score (minimum score = 0, maximum score = 100), the changed ALS non-specific sub-score (minimum score = 0, maximum score = 36), a changed summed total ECAS-N score (minimum score =0, maximum score =136), the changed sub score of behavioural changes (minimum score = 0, maximum score = 10) and the changed sub score of psychotic change (minimum score = 0, maximum score = 3). A changed dichotomized cut-off scores for normality will also be used for the ALS-specific cut-off score of 65 or over, the non ALS-specific cut-off score of 24 or over and the total ECAS-N cut-off score of 92 or over. For the ALS-specific scores, non ALS-specific scores and total ECAS-N scores, high scores indicate less problems than low scores. For the sub score of behavioural change and the sub score of psychotic change, high scores indicate more problems than low scores.
Montreal Cognitive Assessment (MoCA) | 4 months
  We will use the total MoCA score (minimum score = 0, maximum score = 30) and a dichotomized cut-off score for normality of 26 or over. High scores indicate less problems than low scores
Change from 4 months Montreal Cognitive Assessment (MoCA) at 8 months | 8 months
  We will use the changed total MoCA score (minimum score = 0, maximum score = 30) and the changed dichotomized cut-off score for normality of 26 or over. High scores indicate less problems than low scores

CONTACTS AND LOCATIONS:
Overall Officials: Tina Taule, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No